CLINICAL TRIAL: NCT03532802
Title: The Effect of Metoprolol on Myocardial Function, Perfusion, Hemodynamics and Heart Failure Symptoms in Patients With Hypertrophic Obstructive Cardiomyopathy.
Brief Title: The Effect of Metoprolol in Patients With Hypertrophic Obstructive Cardiomyopathy.
Acronym: TEMPO
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Steen Hvitfeldt Poulsen (Other)
Responsible Party: Sponsor-Investigator, Steen Hvitfeldt Poulsen, Senior consultant, DMSc, Aarhus University Hospital, Aarhus University Hospital Skejby
Organization: Aarhus University Hospital Skejby (Other)
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 1-10-72-441-17
Record Dates: First submitted 2018-04-19; First posted 2018-05-22 (Actual); Last update posted 2021-03-29 (Actual); Status verified 2021-03

CONDITIONS: Hypertrophic Cardiomyopathy
Keywords: metoprolol; heart diseases; cardiovascular diseases; ventricular outflow obstruction; hemodynamics
MeSH Terms: conditions — Cardiomyopathy, Hypertrophic; Heart Diseases; Cardiovascular Diseases; Ventricular Outflow Obstruction | interventions — Metoprolol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Metoprolol Succinate (Active Comparator): Metoprololsuccinat
  Interventions: Drug: Metoprolol Succinate
- Placebo oral capsule (Placebo Comparator): Placebo
  Interventions: Drug: Placebo oral capsule

INTERVENTIONS:
Drug: Metoprolol Succinate — 1. week: uptitration with 50 mg capsules per day, until maximum dosage of 150 mg´s/day.
  2. week: steady state treatment with the maximum tolerated dose of the 1.week.
  Arms: Metoprolol Succinate
Drug: Placebo oral capsule — 1. week: uptitration with 1 capsule per day, until maximum tolerated dosage of 3 capsules/day.
  2. week: steady state treatment with the maximum tolerated dose of the 1. week
  Arms: Placebo oral capsule

SUMMARY:
Hypertrophic obstructive cardiomyopathy (HOCM) patients often develop disabling symptoms of heart failure. Current treatment strategies are predicated on the empirical use of long-standing drugs, such as beta-adrenergics, although with little evidence supporting their clinical beneﬁt in this disease. Metoprolol is currently the most widely used beta-blocker in symptomatic HOCM patients, but a randomized, placebo-controlled trial, that looks at the effect in HOCM patients has never been conducted. No studies of HOCM combine invasive pressure measurement with exercise and echocardiography. All previous studies, both invasive and echocardiographic, have been conducted during rest, and not during exercise. Symptoms of HOCM patients are function-related, and exercise testing is essential to assess the condition and the effect of drugs.

DETAILED DESCRIPTION:
Background Hypertrophic cardiomyopathy (HCM) is characterized by an increase in left-ventricular wall thickness, typically localized at the interventricular septum. The hypertrophy can increase to an extend that causes a dynamic obstruction of the left ventricular outflow tract (LVOTO); these patients have hypertrophic obstructive cardiomyopathy (HOCM). Due to the obstruction, patients develop high interventricular pressure gradients, which may overtime become detrimental to the left ventricular function.

HOCM patients often develop disabling symptoms of heart failure. Current treatment strategies are predicated on the empirical use of long-standing drugs, such as beta-adrenergics, although with little evidence supporting their clinical beneﬁt in this disease. Metoprolol is currently the most widely used beta-blocker in symptomatic HOCM patients, but a randomized, placebo-controlled trial, that looks at the effect in HOCM patients has never been conducted. No studies of HOCM combine invasive pressure measurement with exercise and echocardiography. All previous studies, both invasive and echocardiographic, have been conducted during rest, and not during exercise. Symptoms of HOCM patients are function-related, and exercise testing is essential to assess the condition and the effect of drugs.

Objective The investigators wants to quantify the effects of metoprolol on myocardial function and perfusion, hemodynamics and heart failure symptoms in patients with HOCM.

Hypotheses

Primary

• Metoprolol treatment reduces ∆ pulmonary capillary wedge pressure (PCWP) (rest-exercise)

Secondary

* Metoprolol treatment reduces PCWP at rest
* Metoprolol treatment increases maximal oxygen consumption (VO2-max) .
* Metoprolol treatment reduces LVOT gradient during exercise
* Metoprolol treatment increases the coronary flow reserve
* Metoprolol treatment decrease External Work
* Metoprolol treatment reduces heart failure symptoms, estimated by the Kansas City Cardiomyopathy Questionnaire

Design and methods

A randomized, double-blinded, placebo-controlled, crossover study, anticipated to examine 32 patients with HOCM both during treatment with metoprolol and placebo.

Patients will be examined in a set-up of simultaneous 1) right heart catheterization 2) cardiopulmonary exercise test and 3) transthoracic echocardiography. The set-up allows the investigators to evaluate the hemodynamic values during rest and maximum exercise.

ELIGIBILITY:
Inclusion Criteria:

* Wall thickness ≥ 15 mm in one or more myocardial segments that is not explained by loading conditions.
* LVOT gradient > 30 mmHg at rest and/or > 50 mmHg at Valsalva's maneuver or exercise
* New York Heart Association Functional class (NYHA) ≥ II

Exclusion Criteria:

* Age < 18 years
* Known allergy to trial medicine
* Contraindications to beta-blocker treatment
* Contraindications to Magnetic resonans scan, including contraindication to the contrast agent gadolinium.
* Female patients who are pregnant (positive plasma-HCG), breastfeeding or of child-bearing potential while not practicing effective chemical contraceptive hormones.
* In case of patients having a pacemaker, they may not be pace-dependent.
* Treatment with Amiodarone
* Atrial fibrillation/flutter at the time of examination
* Bradycardia < 49 beats/min
* Systolic blood pressure < 100 mmHg
* Trifascicular block
* Previous transcoronary ablation of septum hypertrophy (TASH) or myectomy
* Current abuse of alcohol and/or drugs
* Significant co-morbidity or issues that makes the patient unsuitable for participation, judged by the investigator
* Patients who cannot give valid consent (e.g. mental illness or dementia)
* Patients who do not understand danish

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2020-09-01 (Actual); Study Completion 2020-09-01 (Actual)

PRIMARY OUTCOMES:
∆Pulmonary capillary wedge pressure (rest-exercise) | Changes will be evaluated after an expected average of 2 weeks of treatment in both treatment arms
  Changes in pulmonary capillary wedge pressure in mmHg from rest to exercise, measured during right heart catheterization

SECONDARY OUTCOMES:
Pulmonary capillary wedge pressure at rest | Changes will be evaluated after an expected average of 2 weeks of treatment in both treatment arms
  Changes in pulmonary capillary wedge pressure in mmHg during rest, measured during right heart catheterization
VO2-max | Changes will be evaluated after an expected average of 2 weeks of treatment in both treatment arms
  Changes in maximal oxygen consumption (L/min) measured during cardiopulmonary exercise test
LVOT gradient during maximum exercise | Changes will be evaluated after an expected average of 2 weeks of treatment in both treatment arms
  Changes of the LVOT gradient during maximum exercise, measured in mmHg during 2D echocardiography
Coronary flow reserve | Changes will be evaluated after an expected average of 2 weeks of treatment in both treatment arms
  Changes in the ratio of maximum coronary blood flow (induced by infusion of adenosin) to resting coronary blood flow, estimated by 2D doppler echocardiography
N-terminal prohormone of brain natriuretic peptide | Changes will be evaluated after an expected average of 2 weeks of treatment in both treatment arms
  Changes in level of N-terminal prohormone of brain natriuretic peptide (ng/L) in blood sample
Changes of symptoms and quality of life with Kansas City Cardiomyopathy Questionnaire | Changes will be evaluated after an expected average of 2 weeks of treatment in both treatment arms
  Changes of symptoms and quality of life with Kansas City Cardiomyopathy Questionnaire assessed by clinical evaluation

CONTACTS AND LOCATIONS:
Overall Officials: Steen Hvitfeldt Poulsen, MD, Study Director — Aa; Morten Kvistholm Jensen, MD, PhD, Study Director — Aarhus University Hospital, Department of Cardiology; Torsten Bloch Rasmussen, MD, PhD, Study Director — Aarhus University Hospital, Department of Cardiology
Locations (1):
- Aarhus University Hospital, Department of Cardiology, Aarhus N, Danmark, Denmark

REFERENCES:
- [Derived] Dybro AM, Rasmussen TB, Nielsen RR, Ladefoged BT, Andersen MJ, Jensen MK, Poulsen SH. Effects of Metoprolol on Exercise Hemodynamics in Patients With Obstructive Hypertrophic Cardiomyopathy. J Am Coll Cardiol. 2022 Apr 26;79(16):1565-1575. doi: 10.1016/j.jacc.2022.02.024. PMID 35450573
- [Derived] Dybro AM, Rasmussen TB, Nielsen RR, Andersen MJ, Jensen MK, Poulsen SH. Randomized Trial of Metoprolol in Patients With Obstructive Hypertrophic Cardiomyopathy. J Am Coll Cardiol. 2021 Dec 21;78(25):2505-2517. doi: 10.1016/j.jacc.2021.07.065. PMID 34915981